CLINICAL TRIAL: NCT00332696
Title: Evaluation of the Effect of Octreotide Compared to Placebo in Patients With Inoperable Bowel Obstruction Due to Peritoneal Carcinomatosis
Brief Title: Octreotide Compared to Placebo in Patients With Inoperable Bowel Obstruction Due to Peritoneal Carcinomatosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSMS995AFR08
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Results first posted 2011-06-15 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Peritoneal Neoplasms; Intestinal Obstruction; Carcinomatosis
Keywords: bowel obstruction,; peritoneal carcinomatosis; Octreotide; inoperable
MeSH Terms: conditions — Peritoneal Neoplasms; Intestinal Obstruction; Carcinoma | interventions — Octreotide; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Octreotide (Experimental): Participants received Octreotide long-acting release (LAR) 30 mg intramuscular injection every 28 days for 3 months beginning on Day 1. Participants also received immediate-release Octreotide 600 µg/day (administered subcutaneously 2 or 3 times a day or via continuous intravenous (IV) or subcutaneous injection over a 24 hour period) and methlylpredinisolone 3-4 mg/kg per day (IV bolus for 1 hour or 2 subcutaneous injections) for the first 6 days.
  Interventions: Drug: Octreotide LAR; Drug: Octreotide (Immediate release); Drug: methylprednisolone
- Placebo (Placebo Comparator): Participants received physiologic saline solution intramuscular injection every 28 days for 3 months beginning on Day 1. Participants also received physiologic saline solution (administered subcutaneously 2 or 3 times a day or via continuous intravenous or subcutaneous injection over a 24 hour period) and methlylpredinisolone 3-4 mg/kg per day (IV bolus for 1 hour or 2 subcutaneous injections) for the first 6 days.
  Interventions: Drug: methylprednisolone; Drug: Placebo

INTERVENTIONS:
Drug: Octreotide LAR — Octreotide long-acting release (LAR) 30 mg intramuscular injection.
  Other Names: Sandostatin® LAR
  Arms: Octreotide
Drug: Octreotide (Immediate release) — Immediate-release Octreotide supplied in 100 µg/mL ampules.
  Other Names: Sandostatin®
  Arms: Octreotide
Drug: methylprednisolone — methlylpredinisolone 3-4 mg/kg per day (IV bolus for 1 hour or 2 subcutaneous injections).
Drug: Placebo — Physiologic saline solution
  Arms: Placebo

SUMMARY:
To evaluate in combination with corticosteroid and local standard medical care the efficacy and safety of long-acting octreotide compared to placebo for the treatment of symptoms of inoperable bowel obstruction in patients with peritoneal carcinomatosis

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptoms and signs of inoperable bowel obstruction confirmed by a surgeon or clinic and radiographic assessment (CT scan or at least abdominal X-ray);
* Confirmed peritoneal carcinomatosis (with one of the following criteria : surgery, imaging and/or cytology);
* No corticotherapy at dose more than 1mg/kg equivalent-methylprednisolone, in the previous 2 weeks ;
* No chemotherapy in the previous week;
* No radio or chemotherapy planned at the inclusion and within the two weeks following inclusion
* Authorized concomitant treatments for local standard medical care : antiemetics, antispasmodics, anti-Histamine2 (H2) drugs blockers or proton pump inhibitor, analgesics; nasogastric tube

Exclusion Criteria:

* Abnormal coagulation (prothrombin time < 60%, platelets < 50x10^9/L).
* Non authorized concomitant treatments :

  1. Anticholinergics such as scopolamine
  2. Other somatostatin analogues

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2005-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Créteil, France

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Octreotide | Placebo
Started | 32 | 32
Completed Day 14 Visit | 21 (Primary Endpoint) | 15
Completed | 2 (Completed Month 3 Visit) | 2
Not Completed | 30 | 30
Not completed — Death | 24 | 14
Not completed — Insufficient therapeutic effect | 4 | 11
Not completed — Adverse Event | 1 | 2
Not completed — Condition does not justify treatment | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Octreotide | Placebo | Total
Number analyzed (Participants) | 32 | 32 | 64
Age Continuous [Mean (Standard Deviation); unit: years] | 65.3 (9.57) | 63.1 (12.36) | 64.2 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 21 | 46
  Male | 7 | 11 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Success From Day 10 to Day 13
Description: Treatment Success was defined as: less than 2 episodes of vomiting on average per day for the 4 days prior to Day 14 [from Day 10 to Day 13] and no use of an Nasogastric Tube (NGT) since at least Day 10 and no use of an anticholinergic agent until Day 14.
  Treatment Failure is defined as: 2 or more episodes of vomiting per day on average for the 4 days prior to Day 14 or use of an NGT after Day 9 or use of an anticholinergic agent before Day 14 or withdrawal from the trial between Day 1 and Day 14 (included), whatever the cause.
Time Frame: Day 10 to Day 13
Population: Intent-to-treat population consisted of all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Octreotide | Placebo
Number analyzed (Participants) | 32 | 32
Participants
  TREATMENT SUCCESS | 12 | 9
  Vomiting episodes <2 (per day) | 19 | 13
  Vomiting episodes ≥2 (per day) | 2 | 2
  No Nasogastric Tube since Day 10 | 14 | 13
  Nasogastric Tube used since Day 10 | 7 | 2
  No Anticholinergic agents | 18 | 11
  Anticholinergic agents taken | 3 | 4
  Premature discontinuation/missing data, failure | 11 | 17

2. Secondary Outcome: Number of Participants With Treatment Success From Day 5 to Day 7
Description: Day 7 treatment success was defined as improvement of symptoms in the previous 2 days (average number of vomiting episodes less than 2 from Day 5, no Nasogastric Tube (NGT) since Day 5 and no anticholinergic agent or withdrawal from trial).
Time Frame: Day 5 to Day 7
Population: Intent-to-treat population consisted of all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Octreotide | Placebo
Number analyzed (Participants) | 32 | 32
Participants
  TREATMENT SUCCESS | 22 | 20
  Vomiting episodes <2 (per day) since Day 5 | 28 | 25
  Vomiting episodes ≥2 (per day) since Day 5 | 1 | 2
  No Nasogastric Tube since Day 5 | 22 | 24
  Nasogastric Tube used since Day 5 | 7 | 3
  No Anticholinergic agents | 26 | 25
  Anticholinergic agents taken | 3 | 2
  Premature discontinuation/missing data | 3 | 5

3. Secondary Outcome: Number of Vomiting Episodes Per Day at Day1, Day 2 and Day 14
Description: The mean number of vomiting episodes per a 24 hour period is presented for Day 1, Day 7 and Day 14.
Time Frame: Day 1, Day 7 and Day 14
Population: Intent-to-treat population consisted of all randomized participants who received study drug. "n" in each of the categories is the number of participants with data at the given time point.
Measure: Mean (Standard Deviation); unit: Vomiting episodes
Arm/Group | Octreotide | Placebo
Number analyzed (Participants) | 32 | 32
Vomiting episodes
  Day 1 | 1.2 (2.14) | 0.6 (1.85)
  Day 7 (n=31,31) | 0.3 (0.64) | 0.4 (0.84)
  Day 14 (n=28,27) | 0.3 (0.81) | 0.5 (2.12)

4. Secondary Outcome: Number of Participants Reporting Scores 0 to 3 on the Nausea Intensity World Heath Organization (WHO) Scale at Day 1
Description: Participants rated their nausea intensity on a scale of 0 to 3, with 3 being the worse. The number of participants with a score of 0, a score of 1, a score of 2 and a score of 3 are presented for Day 1.
Time Frame: Day 1
Population: Intent-to-treat population consisted of all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Octreotide | Placebo
Number analyzed (Participants) | 32 | 32
Participants
  Score=0 | 16 | 13
  Score=1 | 1 | 2
  Score=2 | 7 | 9
  Score=3 | 8 | 8

5. Secondary Outcome: Number of Participants Reporting Scores 0 to 3 on the Nausea Intensity World Heath Organization (WHO) Scale at Day 7
Description: Participants rated their nausea intensity on a scale of 0 to 3, with 3 being the worse. The number of participants with a score of 0, a score of 1, a score of 2 and a score of 3 are presented for Day 7.
Time Frame: Day 7
Population: Participants from the Intent-to-treat population consisting of all randomized participants who received study drug and for whom data was available at Day 7.
Measure: Number; unit: Participants
Arm/Group | Octreotide | Placebo
Number analyzed (Participants) | 31 | 31
Participants
  Score=0 | 21 | 15
  Score=1 | 2 | 9
  Score=2 | 5 | 6
  Score=3 | 3 | 1

6. Secondary Outcome: Number of Participants Reporting Scores 0 to 3 on the Nausea Intensity World Heath Organization (WHO) Scale at Day 14
Description: Participants rated their nausea intensity on a scale of 0 to 3, with 3 being the worse. The number of participants with a score of 0, a score of 1, a score of 2 and a score of 3 are presented for Day 14.
Time Frame: Day 14
Population: Participants from the Intent-to-treat population consisting of all randomized participants who received study drug and for whom data was available at Day 14.
Measure: Number; unit: Participants
Arm/Group | Octreotide | Placebo
Number analyzed (Participants) | 28 | 27
Participants
  Score=0 | 22 | 22
  Score=1 | 2 | 3
  Score=2 | 2 | 1
  Score=3 | 2 | 1

7. Secondary Outcome: Number of Participants With Relief From Obstruction at Day 7 and Day 14
Description: Relief from obstruction is defined by combining restart of stools for at least the previous 3 days, less than 2 episodes of vomiting on average for the previous 4 days and the restarting of flatus (gas generated in the stomach or bowels) for at least the previous 12 hours.
Time Frame: Day 7 and Day 14
Population: Intent-to-treat population consisted of all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Octreotide | Placebo
Number analyzed (Participants) | 32 | 32
Participants
  Relief from Obstruction: Day 7 | 9 | 15
  No Relief from Obstruction: Day 7 | 20 | 12
  Relief from Obstruction: Day 14 | 11 | 10
  No Relief from Obstruction: Day 14 | 10 | 5

8. Secondary Outcome: Number of Participants With Recurrence of an Episode of Bowel Obstruction at Month 1
Description: Recurrence of bowel obstruction was confirmed by abdominal X-ray.
Time Frame: 1 Month
Population: Participants from the Intent-to-treat population (consisting of all randomized participants who received at least one dose of study drug) for whom data was available at Month 1.
Measure: Number; unit: Participants
Arm/Group | Octreotide | Placebo
Number analyzed (Participants) | 14 | 15
Participants
  Recurrence at Month 1 | 1 | 2
  No Recurrence at Month 1 | 13 | 13

9. Secondary Outcome: Number of Participants With Recurrence of an Episode of Bowel Obstruction at Month 2
Description: Recurrence of bowel obstruction was confirmed by abdominal X-ray.
Time Frame: Month 2
Population: Participants from the Intent-to-treat population (consisting of all randomized participants who received at least one dose of study drug) for whom data was available at Month 2.
Measure: Number; unit: Participants
Arm/Group | Octreotide | Placebo
Number analyzed (Participants) | 8 | 7
Participants
  Recurrence at Month 2 | 2 | 2
  No Recurrence at Month 2 | 6 | 5

10. Secondary Outcome: Number of Participants With Recurrence of an Episode of Bowel Obstruction at Month 3
Description: Recurrence of bowel obstruction was confirmed by abdominal X-ray.
Time Frame: Month 3
Population: Participants from the Intent-to-treat population (consisting of all randomized participants who received at least one dose of study drug) for whom data was available at Month 3.
Measure: Number; unit: Participants
Arm/Group | Octreotide | Placebo
Number analyzed (Participants) | 3 | 2
Participants
  Recurrence at Month 3 | 0 | 0
  No Recurrence at Month 3 | 3 | 2

11. Secondary Outcome: Participant's Quality of Life Using the Edmonton Scale
Description: The Edmonton Scale consisted of 9 items: pain, activity, nausea, depression, anxiety, fatigue, appetite, sensation of well-being and dyspnea (difficult or labored breathing). Participants rated these items on a scale of 0 to 10, with 10 being the worse.
Time Frame: Day 1, Day 7, Day 14, Month 1, Month 2 and Month 3
Population: Intent-to-treat population consisted of all participants who received at least one dose of study drug. "n" in each of the categories is the number of participants who had Quality of Life data at that time point.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Octreotide | Placebo
Number analyzed (Participants) | 32 | 32
Scores on a scale
  Day 1 (n=30,29) | 4.12 (1.174) | 4.12 (1.360)
  Day 7 (n=24,26) | 4.23 (1.695) | 3.37 (1.247)
  Day 14 (n=20,14) | 4.30 (1.652) | 3.85 (1.860)
  Month 1 (n=11,13) | 4.18 (1.905) | 4.49 (1.820)
  Month 2 (n=7,4) | 3.46 (2.339) | 3.23 (1.609)
  Month 3 (n=2,2) | 0.05 (0.071) | 1.60 (0.283)

ADVERSE EVENTS:
Arm/Group | Octreotide | Placebo
Serious Adverse Events (participants affected / at risk) | 6/32 | 6/32
Other Adverse Events (participants affected / at risk) | 24/32 | 19/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Octreotide (N=32) | Placebo (N=32)
Cardiac arrest (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Disease progression (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 3
Hyperthermia (General disorders) | 1 | 1
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Cytolytic hepatitis (Hepatobiliary disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 2
Septic shock (Infections and infestations) | 1 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Coma (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ileostomy (Surgical and medical procedures) | 0 | 1
Laparotomy (Surgical and medical procedures) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Octreotide (N=32) | Placebo (N=32)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Cardiogenic shock (Cardiac disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 7 | 4
Diarrhoea (Gastrointestinal disorders) | 5 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Melaena (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 7 | 2
Vomiting (Gastrointestinal disorders) | 6 | 5
Asthenia (General disorders) | 7 | 3
Chills (General disorders) | 2 | 0
Condition aggravated (General disorders) | 3 | 1
Disease progression (General disorders) | 7 | 2
Fatigue (General disorders) | 3 | 1
General physical health deterioration (General disorders) | 3 | 3
Hypothermia (General disorders) | 2 | 0
Oedema (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 2 | 3
Pain (General disorders) | 1 | 2
Pyrexia (General disorders) | 3 | 1
Jaundice (Hepatobiliary disorders) | 2 | 1
Oral fungal infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 2
Septic shock (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 3 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Headache (Nervous system disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 3 | 4
Confusional state (Psychiatric disorders) | 4 | 2
Disorientation (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 1
Dysuria (Renal and urinary disorders) | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 3 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Study was terminated prematurely due to low enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure Restriction Description: The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial; or of the trial results in their entirety.